CLINICAL TRIAL: NCT00510159
Title: Randomized Double Blind Clinical Trial in Mali, Comparing the Effectiveness of Artesunate + Sulfamethoxypyrazine/Pyrimethamine Versus Praziquantel in the Treatment of S. Haematobium in Children
Brief Title: Comparing Praziquantel Versus Artesunate + Sulfamethoxypyrazine/Pyrimethamine for Treating Schistosomiasis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Dafra Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2007/S4
Record Dates: First submitted 2007-07-31; First posted 2007-08-01 (Estimated); Last update posted 2008-01-18 (Estimated); Status verified 2007-07

CONDITIONS: Schistosoma Haematobium
Keywords: Schistosoma haematobium; Praziquantel; Artesunate + Sulfamethoxypyrazine/pyrimethamine; Randomized double blind placebo controlled clinical trial
MeSH Terms: conditions — Schistosomiasis haematobia | interventions — Praziquantel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Artesunate+Sulfamethoxypyrazine/pyrimethamin
  Other Names: Co-Arinate FDC ®
Drug: Praziquantel

SUMMARY:
The purpose of this study is to evaluate the efficacy of praziquantel versus As+SMP (Co-Arinate FDC ®) in the treatment of Schistosoma haematobium in 6-15 year old Malian children. The nul-hypothesis in this study is that the combination of As+SMP is more effective than praziquantel in the treatment of S. haematobium infected children.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 6-15 years
* In good health, according to study doctor
* Suffering from urinary schistosomiasis, as diagnosed by the presence of S. haematobium eggs in the urine.
* Residents of Djalakorodji
* Capable of taking oral medication
* Written informed consent to participate in the study, obtained from parent or legal guardian.

Exclusion Criteria:

* Weighing more than 50 kg
* Being pregnant or lactating at the time of the study
* Patient has a severe concomitant disease, as determined by the clinical examination, such as cerebral cysticercosis, HIV,...
* Signs of severe malnutrition (children weighing/measuring more than 3 standard deviations or less than 70% of the median standard reference values determined by WHO, or with systemic oedema affecting both feet).
* Hypersensitivity to As, SMP or PZQ
* Having taken other antimalarial or antischistosomal medication during the study.
* Having participated in previous similar studies

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 800 (Actual)
Dates: Start 2007-08; Primary Completion 2007-10 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Compare the parasite load between the two treatment arms | After 28 days
Compare the amount of eggs produced between the two treatment arms | After 28 days
Compare cure rate between the two treatment arms | After 28 days

SECONDARY OUTCOMES:
Evaluate changes in urine appearance before and after treatment | After 28 days
Evaluate changes in haematuria frequency before and after treatment | After 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Mahamadou S Sissoko, MD, MSPH, Principal Investigator — University of Bamako, Mali
Locations (1):
- Djalakorodji, Mali

REFERENCES:
- [Derived] Sissoko MS, Dabo A, Traore H, Diallo M, Traore B, Konate D, Niare B, Diakite M, Kamate B, Traore A, Bathily A, Tapily A, Toure OB, Cauwenbergh S, Jansen HF, Doumbo OK. Efficacy of artesunate + sulfamethoxypyrazine/pyrimethamine versus praziquantel in the treatment of Schistosoma haematobium in children. PLoS One. 2009 Oct 5;4(10):e6732. doi: 10.1371/journal.pone.0006732. PMID 19802383